CLINICAL TRIAL: NCT04151381
Title: The Effect of Preoperative Aminophylline on the Recovery Profile After Major Pelvi-abdominal Surgeries: Randomized Controlled Double Blinded Study
Brief Title: The Effect of Preoperative Aminophylline
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa Rashwan, Assistant professor of Anesthesiology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Beni-Suef Hospital, operation
Record Dates: First submitted 2019-09-08; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-09

CONDITIONS: Recovery From Anesthesia
MeSH Terms: interventions — Aminophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the control group (Placebo Comparator): the control group (n =15 ) the patients will receive 20 ml of normal saline IV ,20 minutes before induction of general anesthesia .
  Interventions: Drug: Aminophylline
- Amiophylline (2mg) (Active Comparator): Aminophylline 2mg:(n = 15) the patients will receive 2 mg/kg intravenous (IV) aminophylline diluted in 20 ml normal saline 20 minutes before induction of general anesthesia
  Interventions: Drug: Aminophylline
- Aminophylline(4mg) (Active Comparator): Aminophylline 4mg: (n = 15) the patients will receive 4 mg/kg intravenous (IV) aminophylline diluted in 20 ml normal saline 20 minutes before induction of general anesthesia .The study drugs will be given by an anesthetist unaware of the study protocol.
  Interventions: Drug: Aminophylline

INTERVENTIONS:
Drug: Aminophylline — the control group (n =15 ) the patients will receive 20 ml of normal saline IV ,20 minutes before induction of general anesthesia .
  Amiopphylline 2mg:(n = 15) the patients will receive 2 mg/kg intravenous (IV) aminophylline diluted in 20 ml normal saline 20 minutes before induction of general anesthesia .
  Aminophylline 4mg: (n = 15) the patients will receive 4 mg/kg intravenous (IV) aminophylline diluted in 20 ml normal saline 20 minutes before induction of general anesthesia .The study drugs will be given by an anesthetist unaware of the study protocol.

SUMMARY:
Several clinical studies and case reports suggested that aminophylline antagonizes the effects of diazepam , barbiturates , sevoflurane ,morphineand propofol.However, the available results from uncontrolled clinical settings make it difficult to quantify the specific effects of aminophylline on hypnotics and anesthetics

DETAILED DESCRIPTION:
Aminophylline, a theophylline derivative, exerts multiple pharmacological effects, either through phosphodiesterase inhibition (i.e., a potent bronchodilating action, which is often used for the treatment of bronchial asthma) or via adenosine receptor blockade .It is generally considered that the majority of actions ascribed to therapeutic doses of xanthines (caffeine and theophylline) are due to their action as adenosine receptor antagonists.

To the best of the investigator's knowledge this hypothesis was not reported in patients scheduled for major pelvi-abdominal surgeries under general anesthesia , and aminophylline was not given as premedication to test this hypothesis as it was previously administrated after the end of surgery ,also it was recommended by previous clinical studies to evaluate the effective dose of aminophylline that affect the extubation and recovery time.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: 20-60 years
* Males and females patients
* American Society Of Anesthesiology (ASA) physical status I- II .

Exclusion Criteria:

* Patient refusal to participate in this study
* Patient with known sensitivity to aminophylline
* Patients with history of cardiac failure
* Patients with renal or hepatic dysfunction and in chronic alcoholism since clearance of aminophylline is decreased.
* Patients with peptic ulcer, hyperthyroidism, glaucoma,as these conditions may be exacerbated.
* Patients with opioid addiction
* Current treatment with B agonists, anticholinergic agents, tranquilizers, anticonvulsants ,or antidepressants.
* Pregnancy.
* Habitual coffee consumption exceeding 2 cups per day.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
times to lose consciousness( LOC) | from the first second after administration of the anesthetic drugs and for 1-5 minutes
  Times to lose of consciousness( LOC) which is defined as an OAA/S score 2 (loss of responsiveness to light tapping on shoulderor mild shaking with voice command to open eyes)

CONTACTS AND LOCATIONS:
Overall Officials: Samaa ak Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Beni-SuefUniversity, Banī Suwayf
  - Beni-Suef University Hospital, Banī Suwayf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kasim SA, Bahr MH, Abdelkader M, Rashwan DAE. The effect of preoperative aminophylline on the recovery profile after major pelvic-abdominal surgeries: a randomized controlled double-blinded study. BMC Anesthesiol. 2021 Apr 19;21(1):122. doi: 10.1186/s12871-021-01340-7. PMID 33874898